CLINICAL TRIAL: NCT02442375
Title: Uniform FDG-PET Guided GRAdient Dose prEscription to Reduce Late Radiation Toxicity (UPGRADE-RT): a Randomised Controlled Trial With Dose Reduction to the Elective Neck in Head and Neck Squamous Cell Carcinoma
Brief Title: Uniform FDG-PET Guided Gradient Dose Prescription to Reduce Late Radiation Toxicity
Acronym: UPGRADE-RT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: UMC Utrecht (Other); Amsterdam UMC, location VUmc (Other); Maastro Clinic, The Netherlands (Other); Radiotherapiegroep (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UPGRADE-RT v3.5 dd20201201
Record Dates: First submitted 2015-04-21; First posted 2015-05-13 (Estimated); Last update posted 2025-11-18 (Actual); Status verified 2025-10

CONDITIONS: Head and Neck Neoplasms; Carcinoma, Squamous Cell
Keywords: head and neck cancer; accelerated radiotherapy; dose reduction; dose de-escalation; elective lymph nodes; FDG-PET
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Squamous Cell | interventions — Prescriptions

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard dose prescription (Active Comparator): * FDG-PET-scan in treatment mask for radiotherapy planning
  * Accelerated radiotherapy IMRT/VMAT with SIB (34 fraction in 5.5 weeks)
  Interventions: Radiation: standard dose prescription
- FDG-PET guided gradient dose prescription (Experimental): * FDG-PET-scan in treatment mask for radiotherapy planning
  * Accelerated radiotherapy IMRT/VMAT with SIB (34 fraction in 5.5 weeks)
  Interventions: Radiation: FDG-PET guided gradient dose prescription

INTERVENTIONS:
Radiation: standard dose prescription — * standard elective dose
  * no intermediate dose-level
  * visual interpretation of FDG-PET-scan
  Arms: standard dose prescription
Radiation: FDG-PET guided gradient dose prescription — * de-escalation of elective dose
  * intermediate dose-level
  * standardized methods to evaluate FDG-PET-scan
  Arms: FDG-PET guided gradient dose prescription

SUMMARY:
The objective of the UPGRADE-RT trial is to investigate whether de-escalation of elective radiation dose and introduction of an intermediate dose-level in the treatment of head and neck cancer will results in less radiation sequelae and improved quality of life after treatment whilst the recurrence rate in electively irradiated lymph nodes should not be compromised.

The full study protocol can be found here:

https://doi.org/10.1200/jco-24-02194

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed tumours classified as stage T2-4 N0-2 (TNM 7th edition 2009) located in the larynx, oropharynx or hypopharynx (unknown primary and oral cavity are not eligible)
2. Histopathological diagnosis of invasive squamous cell carcinoma in the primary tumour
3. Decision for curative intent external beam radiotherapy with elective treatment of the neck made by a multidisciplinary head-and-neck oncology team. The patient must be expected to complete the treatment.
4. Radiotherapy planned to start within 6 weeks from baseline imaging of tumour assessment
5. No distant metastasis (M0) (TNM 7th edition 2009)
6. WHO performance status 0-2
7. ≥ 18 years of age
8. Written informed consent

Exclusion Criteria:

1. Concomitant chemotherapy or EGFR inhibitors for this tumour.
2. Primary tumour of the oral cavity or unknown primary tumour
3. Prior or current anticancer treatment to the head and neck area (e.g. radical attempted or tumour reductive surgery, neo-adjuvant or concomitant chemotherapy, EGFR inhibitors or radiotherapy), except for endoscopic glottic laser micro surgery.
4. Current participation in any other oncologic interventional clinical study for this tumor.
5. Uncontrolled diabetes mellitus.
6. Known or suspected HIV infection.
7. History of previous malignancy within the last 3 years, with the exception of surgically cured carcinoma in situ of the cervix, in situ breast cancer, incidental finding of stage T1a or T1b prostate cancer, basal/squamous cell carcinoma of the skin, and other non-invasive malignancies (e.g. in situ carcinomas)..
8. Any condition (somatic, psychological, familial, sociological or geographical) rendering the patient unable to understand or complete questionnaires.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2024-07-03 (Actual); Study Completion 2024-07-03 (Actual)

PRIMARY OUTCOMES:
Toxicity: normalcy of diet (score of the performance status scale for head and neck cancer patients) | 12 months

SECONDARY OUTCOMES:
Safety: recurrence in electively irradiated lymph nodes | 24 months
  A Kaplan-Meier estimate will be calculated

OTHER OUTCOMES:
Acute toxicity (common toxicity criteria v2.0) | up to 3 months
Late toxicity: swallowing function (water swallowing test) | 3, 12 and 24 months
Late toxicity: salivary gland function (stimulated flow rates) | 3, 12 and 24 months
Late toxicity: thyroid gland function (thyroid stimulating hormone blood test) | 3, 12 and 24 months
Quality of life (EORTC QLQ-C30 and QLQ-H&N35 questionnaires) | 3, 6, 12 and 24 months
Xerostomia related quality of life (GRIX questionnaire) | 3, 6, 12 and 24 months
Dysphagia related quality of life (SWAL-QOL questionnaire) | 3, 6, 12 and 24 months
Loco-regional control | 24 months
  A Kaplan-Meier estimate will be calculated
Overall survival | 24 months
  A Kaplan-Meier estimate will be calculated
Disease specific survival | 24 months
  A Kaplan-Meier estimate will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. J.H.A.M. Kaanders, Study Chair — Radboud University Nijmegen Medical Center
Locations (5):
- Netherlands (5):
  - VU University Medical Center Amsterdam, Amsterdam
  - Radiotherapiegroep, Arnhem, Arnhem
  - MAASTRO clinic, Maastricht, Maastricht
  - Radboud University Nijmegen Medical Center, Nijmegen
  - University Medical Center Utrecht, Utrecht

REFERENCES:
- [Result] van den Bosch S, Doornaert PAH, Hoebers FJP, Kreike B, Vergeer MR, Zwijnenburg EM, Cox MC, Hannink G, Dijkema T, Kaanders JHAM; Dutch Head and Neck Society. Clinical Benefit and Safety of Reduced Elective Dose in Definitive Radiotherapy for Head and Neck Squamous Cell Carcinoma: The UPGRADE-RT Multicenter Randomized Controlled Trial. J Clin Oncol. 2025 Aug 10;43(23):2583-2594. doi: 10.1200/JCO-24-02194. Epub 2025 Apr 15. PMID 40233286
- [Result] van den Bosch S, Cox MC, Doornaert PAH, Hoebers FJP, Kreike B, Vergeer MR, Zwijnenburg EM, Hannink G, Dijkema T, Kaanders JHAM; Dutch Head and Neck Society. Dose de-escalation of elective neck irradiation in head and neck cancer: A secondary analysis of acute toxicity findings from the randomized controlled UPGRADE-RT trial. Radiother Oncol. 2025 Dec;213:111196. doi: 10.1016/j.radonc.2025.111196. Epub 2025 Oct 5. PMID 41057084
- [Derived] van den Bosch S, Dijkema T, Kunze-Busch MC, Terhaard CH, Raaijmakers CP, Doornaert PA, Hoebers FJ, Vergeer MR, Kreike B, Wijers OB, Oyen WJ, Kaanders JH. Uniform FDG-PET guided GRAdient Dose prEscription to reduce late Radiation Toxicity (UPGRADE-RT): study protocol for a randomized clinical trial with dose reduction to the elective neck in head and neck squamous cell carcinoma. BMC Cancer. 2017 Mar 21;17(1):208. doi: 10.1186/s12885-017-3195-7. PMID 28327089